CLINICAL TRIAL: NCT06402760
Title: A Cohort Study on Comprehensive Intervention of Diabetes and Psoriasis Comorbidity Prevention and Control Using Traditional Chinese Medicine of Blood-activating and Stasis-dissolving Method
Brief Title: Comprehensive Intervention of Diabetes and Psoriasis Comorbidity Prevention and Control
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shanghai Hongkou District Center for Disease Control And Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GWVI-11.1-24
Record Dates: First submitted 2024-04-09; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis; Diabetes
MeSH Terms: conditions — Psoriasis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Western medicine group (Active Comparator): Treatment will be stratified according to the severity of psoriasis in patients, with therapeutic methods limited to the traditional treatment approaches outlined in the Chinese Guidelines for the Diagnosis and Treatment of Psoriasis (2023 Simplified Version). The treatment duration will be 16 weeks, followed by a 24-week follow-up period during which patients will not be restricted in their treatment modalities.
  Interventions: Drug: Western medicine
- TCM comprehensive treatment group (Experimental): In addition to the Western medicine treatment prescribed in the guidelines, patients are required to take fish oil orally and Taodan Granules, and engage in moderate to high-intensity aerobic exercise weekly.
  Interventions: Other: TCM comprehensive treatment

INTERVENTIONS:
Other: TCM comprehensive treatment — 1. Taodan Granules (TCM formulation for promoting blood circulation and removing blood stasis): The granules consist of the following herbal components: milkvetch, licorice, angelica, rhizoma chuanxiong, peach seed, Salvia miltiorrhiza, Curcuma zedoaria, Achyranthes bidentata, and sarsaparilla. Patients will take it orally in two divided doses after breakfast and dinner.
  2. Fish Oil: Patients will take 1g of fish oil orally twice daily. Patients will be instructed to purchase fish oil under the guidance of the researchers.
  3. Exercise Plan: Researchers will design an exercise plan for patients, who will be required to engage in at least 150 minutes of moderate-intensity aerobic exercise per week.
  Patients will undergo a 16-week treatment period followed by a 24-week follow-up period. During the follow-up, patients will continue taking fish oil and adhering to the exercise regimen, while other treatment modalities will be unrestricted.
  Arms: TCM comprehensive treatment group
Drug: Western medicine — The treatment methods prescribed in the guidelines.
  Arms: Western medicine group

SUMMARY:
We will recruit 300 patients with psoriasis from Yueyang Hospital of Integrative Medicine, Shanghai University of Traditional Chinese Medicine, who will not be currently diagnosed with diabetes but will have been identified as high-risk individuals based on the developed risk assessment model. Based on doctor's treatment opinions and patient preferences, participants will be divided into two groups in a 1:1 ratio: a Western medicine group and a TCM comprehensive treatment group.

Patients in the Western medicine group will receive treatment according to guidelines. Patients in the TCM comprehensive treatment group will be treated according to the guidelines and will additionally receive Taodan granules (to be taken daily during the treatment period after brewing the granules with lukewarm water in the morning and evening) and fish oil (1g, taken orally twice daily).

Patients in the TCM comprehensive treatment group will be required to complete at least 150 minutes of moderate-intensity aerobic exercise per week under the supervision of a physician. The patients will be treated for 16 weeks and followed up for 24 weeks to see if the treatment prevents the development of diabetes or insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Western medicine diagnostic criteria for vulgaris psoriasis and the Traditional Chinese Medicine diagnostic criteria for blood stasis syndrome in psoriasis.
2. Newly diagnosed or previously diagnosed with psoriasis; if previously diagnosed, prior treatment methods are not restricted.
3. Identified as high risk for comorbid diabetes based on a risk model calculation.
4. Age between 18 and 80 years old, any gender.
5. Willing to participate in this study and provide informed consent.

Exclusion Criteria:

1. Patients already diagnosed with diabetes.
2. Presence of other active skin diseases that may affect the assessment of the condition.
3. In severe, difficult-to-control acute or chronic infection locally or systemically.
4. Severe systemic diseases; or patients with clinical laboratory indicators falling into any of the following conditions:

   ① Hematology: Hemoglobin (HGB) < 90g/L; Platelet count (PLT) < 10010^9/L; White blood cell count (WBC) < 310^9/L; Absolute neutrophil count (NEUT) < 1.5*10^9/L;

   ② Liver function: Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) exceeding 3 times the upper limit of normal (ULN) or total bilirubin exceeding 1.5 times the upper limit of normal;

   ③ Renal function: Serum creatinine greater than 1.5 times the upper limit of normal;

   ④ Other abnormal laboratory test results judged by the investigator to potentially affect the patient's completion of the trial or interfere with the trial results.
5. History of malignant tumors and primary or secondary immunodeficiency or hypersensitivity.
6. Underwent major surgery within 8 weeks or will require such surgery during the study period.
7. Pregnant or lactating women.
8. History of alcoholism, drug abuse, or substance abuse.
9. History of severe mental illness or family history thereof.
10. Family history of tumors.
11. Other reasons deemed inappropriate for participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of participants assessed for diabetes prevention efficacy based on Glycated Hemoglobin (HbA1c) | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40)
  The members of the two groups will measure glycosylated hemoglobin (HbA1c) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine at the 16th week of treatment and the follow-up period (40th week) to judge whether diabetes or insulin resistance occurs.
The number of participants assessed for diabetes prevention efficacy based on Fasting Plasma Glucose (FPG) | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40)
  The members of the two groups will measure Fasting Plasma Glucose (FPG) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine at the 16th week of treatment and the follow-up period (40th week) to judge whether diabetes or insulin resistance occurs.
The number of participants assessed for diabetes prevention efficacy based on Postprandial 2-hour Plasma Glucose (PPG) | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40)
  The members of the two groups will measure Plasma Glucose (PPG) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine at the 16th week of treatment and the follow-up period (40th week) to judge whether diabetes or insulin resistance occurs.
The number of participants assessed for diabetes prevention efficacy based on Fasting Insulin (FINS) | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40)
  The members of the two groups will measure Fasting Insulin (FINS) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine at the 16th week of treatment and the follow-up period (40th week) to judge whether diabetes or insulin resistance occurs.
The number of participants assessed for diabetes prevention efficacy based on C-peptide | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40)
  The members of the two groups will measure C-peptide in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine at the 16th week of treatment and the follow-up period (40th week) to judge whether diabetes or insulin resistance occurs.
The number of participants assessed for psoriasis improvement efficacy due to clinical intervention based on Improvement of PASI (Psoriasis Area and Severity Index). | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40)
  Improvement of PASI= PASI at week 0 - PASI at week 16 and week 40.

SECONDARY OUTCOMES:
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on serum triglyceride (TG) evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will test the serum triglyceride (TG) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on Serum Total Cholesterol (TC) evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will test the Serum Total Cholesterol (TC) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on erum High-Density Lipoprotein Cholesterol (HDL) evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will test the Serum High-Density Lipoprotein Cholesterol (HDL) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on Serum Low-Density Lipoprotein Cholesterol (LDL) evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will test the Serum Low-Density Lipoprotein Cholesterol (LDL) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on Serum Apolipoprotein AI (ApoAI) evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will test Serum Apolipoprotein AI (ApoAI) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on Serum Apolipoprotein B (ApoB) evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will test Serum Apolipoprotein B (ApoB) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on Serum Lipoprotein α evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will test Serum Lipoprotein α in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
The number of participants assessed for improvement in metabolic indicators related to comorbid psoriasis and diabetes due to clinical intervention based on Serum small dense low-density lipoprotein (sdLDL) evaluation. | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of the two groups will testSerum small dense low-density lipoprotein (sdLDL) in Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine to determine whether the metabolic situation related to psoriasis and diabetes is improving.
Assessing the number of participants experiencing a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes using HsCRP | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of both groups will undergo HsCRP testing at the Yueyang Integrative Medicine Hospital affiliated with Shanghai University of Traditional Chinese Medicine to assess whether there is a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes.
Assessing the number of participants experiencing a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes using IL-1β | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of both groups will undergo IL-1β testing at the Yueyang Integrative Medicine Hospital affiliated with Shanghai University of Traditional Chinese Medicine to assess whether there is a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes.
Assessing the number of participants experiencing a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes using IL-6 | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of both groups will undergo IL-6 testing at the Yueyang Integrative Medicine Hospital affiliated with Shanghai University of Traditional Chinese Medicine to assess whether there is a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes.
Assessing the number of participants experiencing a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes using TNFα | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of both groups will undergo TNFα testing at the Yueyang Integrative Medicine Hospital affiliated with Shanghai University of Traditional Chinese Medicine to assess whether there is a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes.
Assessing the number of participants experiencing a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes using IL-17A | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of both groups will undergo IL-17A testing at the Yueyang Integrative Medicine Hospital affiliated with Shanghai University of Traditional Chinese Medicine to assess whether there is a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes.
Assessing the number of participants experiencing a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes using FGL1 | Assessed at screening (Week 0), Week 16 of treatment, and during follow-up (Week 40).
  The members of both groups will undergo FGL1 testing at the Yueyang Integrative Medicine Hospital affiliated with Shanghai University of Traditional Chinese Medicine to assess whether there is a decrease in levels of inflammatory biomarkers associated with the comorbidity of psoriasis and diabetes.
The number of participants assessed for psoriasis improvement efficacy due to clinical intervention based on Improvement of Body Surface Area (BSA). | Assessed at screening (Week 0), Week 4, Week 8, Week 12, Week 16 of treatment, and during follow-up (Week 20, Week 24, Week 28, Week 32, Week 36, Week 40).
  The percentage of BSA involved in psoriasis is estimated by the handprint method, in which the patient's entire palm (that is, the patient's fully outstretched palm, fingers, and thumb) represents about 1% of the total BSA
The number of participants assessed for psoriasis improvement efficacy due to clinical intervention based on Improvement of Physician's Global Assessment (PGA). | Assessed at screening (Week 0), Week 4, Week 8, Week 12, Week 16 of treatment, and during follow-up (Week 20, Week 24, Week 28, Week 32, Week 36, Week 40).
  The PGA is a 5-point scale that is used to reflect the overall assessment of erythema (E), infiltration (I), and desquamation (D) in psoriatic lesions.
The number of participants assessed for psoriasis improvement efficacy due to clinical intervention based on Improvement of Dermatology Life Quality Index (DLQI). | Assessed at screening (Week 0), Week 4, Week 8, Week 12, Week 16 of treatment, and during follow-up (Week 20, Week 24, Week 28, Week 32, Week 36, Week 40).
  The DLQI is a 10item questionnaire assessing the impact of skin disease on health-related quality of life (HRQOL). The total score ranges from 0 to 30; higher scores indicate a lower quality of life . Foreign clinical studies have reported that its 4 Evidence-Based Complementary and Alternative Medicin
  minimal clinically important difference (MCID) is 5 points [30]. +at is, after treatment, DLQI is decreased by 5 points, which can be considered an improvement in quality of life and treatment efficacy.
The number of participants assessed for psoriasis improvement efficacy due to clinical intervention based on Improvement of Psoriasis-related Quality of Life (PRQoL). | Assessed at screening (Week 0), Week 4, Week 8, Week 12, Week 16 of treatment, and during follow-up (Week 20, Week 24, Week 28, Week 32, Week 36, Week 40).
  The questionnaire consists of 15 questions, including five parts: daily activities, at work, personal relationships, leisure activities, and treatment. +e answer to each question gives a score from 0 to 3. +e choice of each question is "very many" (3 points), "a lot" (2 points), "a little" (1 point), and "no answer at all" (0 points)
The number of participants assessed for psoriasis improvement efficacy due to clinical intervention based on Improvement of self-assessment of itching symptoms (VAS) score. | Assessed at screening (Week 0), Week 4, Week 8, Week 12, Week 16 of treatment, and during follow-up (Week 20, Week 24, Week 28, Week 32, Week 36, Week 40).
  VAS is an often-used tool to measure subjective phenomena, which has shown good reliability and validity in terms of assessment of pain. In the clinical study of psoriasis, it can be used as a tool to measure the degree of pruritus from 0 to 100 mm (with 0 being no pruritis and 100 being maximum pruritis).
The number of participants assessed for psoriasis improvement efficacy due to clinical intervention based on Improvement of Traditional Chinese Medicine symptom score. | Assessed at screening (Week 0), Week 4, Week 8, Week 12, Week 16 of treatment, and during follow-up (Week 20, Week 24, Week 28, Week 32, Week 36, Week 40).
  Traditional Chinese Medicine symptom score is used to assess changes in syndrome-related symptoms during treatment.

IPD SHARING:
Plan to Share IPD: No